CLINICAL TRIAL: NCT00017550
Title: An Open Label, Prospective, Stratified, Randomized, Controlled, Multi-Center, Phase IIB Study of the Impact of Thymoglobulin Therapy on Transfusion Needs of Patients With Early Myelodysplastic Syndrome (MDS)
Brief Title: Antithymocyte Globulin Compared With Supportive Care in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Organization: Sanofi (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068709; SMC-101-1020; RUSH-MDS-2000-04
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2003-03

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with excess blasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — Antilymphocyte Serum

INTERVENTIONS:
Biological: anti-thymocyte globulin

SUMMARY:
RATIONALE: Immunosuppressive therapy may improve bone marrow abnormalities and may be effective treatment for myelodysplastic syndrome. It is not yet known whether immunosuppressive therapy is more effective than supportive care in treating myelodysplastic syndrome.

PURPOSE: Randomized phase II trial to compare the effectiveness of antithymocyte globulin with that of supportive care in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the clinical response rate of patients with early myelodysplastic syndrome treated with rabbit anti-thymocyte globulin vs standard supportive care.
* Evaluate the safety of anti-thymocyte globulin in these patients.
* Compare the time to and duration of clinical response, rates of partial response and therapy failure, and rate of disease progression in patients treated with these regimens.
* Compare the ECOG performance score, number of transfusions and/or growth factor use, and maximum time between transfusions in patients treated with these regimens.
* Compare the infection risk, use of medical resources, and quality of clinical response in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to myelodysplastic syndrome (MDS) subtype (refractory anemia (RA) vs RA with excess blasts or hypocellular MDS). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive rabbit anti-thymocyte globulin (ATG) IV over at least 8-12 hours on days 1-4.
* Arm II: Patients receive standard supportive therapy for 6 months. At the end of 6 months, patients may receive ATG as in arm I.

Patients are followed for 6 months.

PROJECTED ACCRUAL: A total of 72 patients (48 in arm I and 24 in arm II) will be accrued within a minimum of 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed early myelodysplastic syndrome (MDS) with less than 10% bone marrow blasts

  * Refractory anemia (RA)
  * RA with excess blasts (RAEB)
  * Hypocellular myelodysplasia
* Low or intermediate-1 prognostic risk
* Transfusion-dependent

  * Need for 2 or more units of red blood cells or platelets per month for 2 or more months prior to study OR
  * History of prior transfusions and 2 consecutive (at least 21 days apart) hemoglobin levels less than 8.0 g/dL or platelet counts less than 20,000/mm^3 during the past 2 months

    * Hemoglobin no greater than 12.0 g/dL after prior transfusion
* No myelosclerosis occupying more than 30% of bone marrow space
* No RA with ringed sideroblasts, RAEB in transformation, or chronic myelomonocytic leukemia
* No therapy-related MDS
* No history of immune-related hematologic disorder (e.g., idiopathic thrombocytopenic purpura)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* See Disease Characteristics
* No other causes of cytopenia unrelated to MDS (e.g., gastrointestinal blood loss)
* Iron present on marrow examination OR
* Transferrin saturation at least 20% and ferritin at least 50 ng/mL

Hepatic:

* Bilirubin no greater than 2 mg/dL OR
* SGOT/SGPT no greater than 2 times normal
* No active or chronic hepatitis B or C

Renal:

* Creatinine no greater than 2 mg/dL

Cardiovascular:

* No symptomatic cardiac disease
* No congestive heart failure (even if medically controlled)
* No myocardial infarction within the past 6 months

Pulmonary:

* No severe pulmonary disease
* If history of pulmonary insufficiency, must have pO_2 at least 90 mm/Hg on room air or pCO_2 no greater than 40 mm/Hg

Other:

* No history of unresolved B12 or folate deficiency since diagnosis of MDS
* No untreated acute or chronic infection (afebrile for 7 days without antibiotics prior to study)
* No active or chronic HIV
* No concurrent cytomegalovirus infection
* No other malignancy within the past 2 years except adequately treated localized squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No concurrent drug or alcohol abuse
* No significant medical or psychosocial problems
* No known allergy to rabbit protein
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 8 weeks since prior biologic agents, colony-stimulating factors, or epoetin alfa for MDS
* At least 8 weeks since other prior investigational biologic agents
* No prior or concurrent bone marrow transplantation
* No concurrent epoetin alfa
* No concurrent growth factors except filgrastim (G-CSF) or sargramostim (GM-CSF) for neutropenic fevers
* No other concurrent biologic agents

Chemotherapy:

* At least 8 weeks since prior cytotoxic drugs for MDS
* Concurrent chemotherapy for clinical indications of disease progression or leukemic transformation allowed

Endocrine therapy:

* At least 8 weeks since prior androgenic hormonal therapy for MDS
* At least 8 weeks since prior danazol for MDS

Radiotherapy:

* No prior radiotherapy

Surgery:

* No prior organ transplantation

Other:

* At least 8 weeks since prior investigational drugs
* At least 8 weeks since prior immunosuppressive drugs or other drugs for MDS
* No concurrent immunosuppressive therapy
* No other concurrent experimental drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09 (Actual); Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C. Squiers, MD, Study Chair — Sangstat Medical Corporation
Locations (28):
- United States (25):
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - University of Florida Health Science Center, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Tampa (Haley), Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Rush Cancer Institute, Chicago, Illinois
  - Indiana Blood and Marrow Transplant, Beech Grove, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Missouri Kansas City School of Medicine, Kansas City, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Texas Oncology P.A., Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Foothills Hospital, Calgary, Alberta
  - Department of Medicine, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario